CLINICAL TRIAL: NCT01415687
Title: A Randomized Prospective Trial Comparing Pico-Salax (Magnesium Citrate) Plus Bisacodyl Versus Split Dose Polyethylene Glycol-Based Lavage In Preparation Of Patients For Colonoscopy
Brief Title: Split Dose Pico-Salax + Bisacodyl vs. PEG Split Dose
Acronym: BP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Alaa Rostom, MD MSc FRCPC, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 23798
Record Dates: First submitted 2011-08-05; First posted 2011-08-12 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: preoperative care; colonoscopy; cathartics
MeSH Terms: interventions — Golytely; Pico-Salax; magnesium citrate; Bisacodyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG Arm (Active Comparator): Patients randomized to this arm of the trial will be following preparation instructions using Polyethylene Glycol-Based Lavage in a split dose format
  Interventions: Drug: Polyethylene Glycol-Based Lavage
- Pico-Salax + Bisacodyl Arm (Active Comparator): Patients randomized to this arm will follow preparation instructions using Pico-Salax preparation plus Biscacodyl in a split dose format
  Interventions: Drug: Pico-Salax (Magnesium Citrate) plus Bisacodyl

INTERVENTIONS:
Drug: Polyethylene Glycol-Based Lavage — Split dose Polyethylene Glycol-Based Lavage (2L + 2L)
  If arrival for colonoscopy is prior to 10AM: at 12 noon on the day before your colonoscopy drink 2L of PEG within two hours. At 8PM that day, drink the remaining 2L of PEG within two hours.
  If arrival for colonoscopy is at or after 10AM: at 8PM on the day before your colonoscopy, drink 2L of PEG within two hours. Starting five hours before your arrival time at the Centre on the day of your colonoscopy, drink the remaining 2L of PEG within two hours.
  Other Names: Colyte
  Arms: PEG Arm
Drug: Pico-Salax (Magnesium Citrate) plus Bisacodyl — If arrival for colonoscopy is prior to 10AM: 2 tablets Dulcolax at 8PM three days before colonoscopy, 2 tablets Dulcolax at 8PM two days before colonoscopy, and on the day before colonoscopy at 12 noon, drink the first packet of Pico-Salax in 8oz water, and the second packet of Pico-Salax in 8oz of water at 8PM. Day of colonoscopy, drink clear fluids.
  If arrival for colonoscopy is at or after 10AM: 2 tablets Dulcolax at 8PM three days before colonoscopy, 2 tablets Dulcolax at 8PM two days before colonoscopy, and on the day before colonoscopy at 8PM, drink the first packet of Pico-Salax in 8oz water. Day of colonoscopy, drink the second packet of Pico-Salax in 8oz water five hours before you are to arrive at the Centre.
  Other Names: Pico-Salax or Magnesium Citrate; Bisacodyl is also known as Dulcolax.
  Arms: Pico-Salax + Bisacodyl Arm

SUMMARY:
The objective of this study is to compare the efficacy, safety and tolerability of two bowel preparations for colonoscopy - split dose Polyethylene Glycol-Based Lavage and Pico-Salax plus Bisacodyl - with a specific emphasis on the right colon cleanliness.

The primary outcomes will be 1) quality of preparation in cleansing the colon, 2) quality of preparation in cleansing the right colon, 3) patient satisfaction. The secondary outcomes will be 1) duration of bowel preparation, 2) patient discomfort during bowel preparation.

DETAILED DESCRIPTION:
All patients referred to the Forzani MacPhail Colon Cancer Screening Centre (CCSC) in Calgary, Alberta, Canada for colonoscopy will be considered for inclusion. During pre-assessments at the clinic, patients are asked to consider a general research consent. If they agree to that, then they will be approached for consideration of participating in this study and presented with an "Invitation to Participate in a Research Study" form (appendix); the study assistant will obtain final consent if they agree. Those not interested in participating will simply receive their physician's standard bowel preparation protocol. There will be no coercion of any sort. Enrollment of participants will be performed with block randomizations of 8 by using a computer-generated table, with allocation concealment maintained through the use of consecutively numbered sealed envelopes. Colonoscopists and investigators will be blinded to allocation groups. Patients will be allocated to one of two groups: (1) oral Pico-Salax (two sachets, with 1.5-2L of water following each sachet) with Dulcolax (Bisacodyl, 4 tablets); (2) split dose Polyethylene Glycol-Based Lavage (2L + 2L).

A study assistant will assign patients to their group and instruct them on the proper use of their assigned bowel preparation method. Patients will be given a tolerability questionnaire, which has been modified from a previously used questionnaire, to be completed once their bowel preparation is finished and before coming to the CCSC for the colonoscopy (included in the appendix). Patient concerns or questions regarding the preparation will be directed toward the study assistant or clinic nurses as opposed to their endoscopist, so as to avoid un-blinding the Colonoscopist. The physician performing the procedure will then complete an Ottawa Bowel Preparation Scale and a validated Simplified Bowel Preparation scale to assess colon cleanliness.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 74 years referred to the in Calgary, Alberta, Canada for colonoscopy will be considered for inclusion

Exclusion Criteria:

* Any history of kidney problems

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quality of Bowel Cleanliness | Scales provided to physician at time of colonoscopy, and filled out and collected after procedure is completed (1 hour time). Questionnaires are manually entered by an assistant into the study database on the same day as collection.
  Ottawa bowel Prep scale will be done by the Dr. to assess the quality of bowel cleanliness. The right, mid and rectosigmoid colon are each rated on a 5-point scale (0-4). Also, a complete 3-point rating for overall colonic fluid is assessed giving an overall score range of 0-14. An excellent preparation would score 0-1; a good preparation, 2-4; while scores >4 would indicate progressively worsening bowel preparations. A completely unprepared colon would score 11-14, depending on the amount of fluid. A simplified overall cleanliness score will be completed and compared to the Ottawa scale.

SECONDARY OUTCOMES:
Patient Satisfaction with preparation | Questionnaire given on day of pre-screen and collected on day of colonoscopy, approximately 3 weeks.Patients are not followed or contacted past the day of colonoscopy.
  Patients will be given an anonymous tolerability questionnaire, which has been modified from a previously used questionnaire, to be completed once their bowel preparation is finished and before coming to the Centre for the colonoscopy. The tool asks questions of patient satisfaction with preparation, ease or difficulty of completing satisfaction, and side effects of the preparation method used.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Rostom, MD, Principal Investigator — University of Calgary Faculty of Medicine
Locations (2):
- Canada (2):
  - Foranzi & MacPhail Colon Cancer Screening Centre, Alberta Health Services, Calgary, Alberta
  - Foranzi & MacPhail Colon Cancer Screening Centre, Calgary, Alberta

REFERENCES:
- [Derived] Rostom A, Dube C, Bishay K, Antonova L, Heitman SJ, Hilsden R. A randomized clinical prospective trial comparing split-dose picosulfate/ magnesium citrate and polyethylene glycol for colonoscopy preparation. PLoS One. 2019 Mar 28;14(3):e0211136. doi: 10.1371/journal.pone.0211136. eCollection 2019. PMID 30921345